CLINICAL TRIAL: NCT06566053
Title: Establishment of a Predictive System for Perioperative Risk Assessment and Electronic Flowcharting Response Strategies in Thoracic Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Hengxing Liang (Other)
Collaborators: Changsha Xinghong Network Technology Co. (Unknown)
Responsible Party: Sponsor-Investigator, Hengxing Liang, Associate professor, Central South University
Organization: Central South University (Other)
Other Study IDs: LYF2023105
Record Dates: First submitted 2024-05-26; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Perioperative Complications
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent thoracic surgery: Gender:Both Participant age:18-100 Examples include early-stage non-small cell lung cancer (NSCLC), NSCLC patients who have undergone neoadjuvant therapy, esophageal diseases, mediastinal masses, chest wall disorders, and other related conditions.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
1. To establish a risk assessment scale for thoracic surgery for the Chinese population, and to classify patients; risk according to the relevant scale;
2. Combining the guidelines for the management of acute and critical illnesses in thoracic surgical care units and the characteristics of diagnosis and treatment operations, to make an AI-assisted diagnosis and treatment process software;
3. Evaluate whether the software can provide timely and correct diagnosis and treatment recommendations for critically ill patients, shorten the time for homogenized training of specialist intensivists, and reduce the hospitalization cost of patients under the review of resident training instructors of various specialties.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Department of Thoracic Surgery of the Second Xiangya Hospital of Central South University for surgical treatment.

Exclusion Criteria:

* Patients admitted to the Department of Thoracic Surgery of the Second Xiangya Hospital of Central South University without surgical treatment.

Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Thoracic Surgery of the Second Xiangya Hospital of Central South University for surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Acute Respiratory Distress Syndrome | 2024.8-2024.12
  ARDS definition was based on the new global definition of ARDS10. Briefly, intubated ARDS was defined as an oxygenation index of less than 300 under a positive end-expiratory pressure (PEEP) of at least 5 cmH2O, and non-intubated ARDS was defined as patients receiving high-flow nasal oxygen (HFNO) ≥ 30 L/min or noninvasive ventilation/continuous positive airway pressure (NIV/CPAP) with a PEEP of at least 5 cmH2O and meeting PaO2:FiO2 ≤ 300 mm Hg or SpO2:FiO2 ≤ 315 (if SpO2 ≤ 97%).

SECONDARY OUTCOMES:
In hospital mortality | 2024.8-2024.12
  refers to the number or percentage of patients who die while being treated in a hospital.
Length of hospital stay | 2024.8-2024.12
  Length of hospital stay(days): refers to the total number of days a patient spends in the hospital from the time of admission to the time of discharge.
Length of ICU stay | 2024.8-2024.12
  Length of ICU stay(hours): refers to the total duration of time a patient spends in the Intensive Care Unit (ICU) during a single admission.
Length of postoperative stay | 2024.8-2024.12
  Length of postoperative stay(days): refers to the duration of time a patient remains in the hospital or medical facility after undergoing surgery.
Duration of mechanical ventilation | 2024.8-2024.12
  Duration of mechanical ventilation(hours): refers to the length of time a patient requires assistance from a mechanical ventilator to maintain adequate breathing.
Duration of HFNC | 2024.8-2024.12
  Duration of HFNC(hours): refers to the length of time that a patient is treated with High-Flow Nasal Cannula (HFNC) therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes